CLINICAL TRIAL: NCT03194477
Title: Identifying and Engaging Urban HIV Infected and Uninfected YBMSM in Care
Brief Title: Providing Unique Support for Health (PUSH) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01DA04308901
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: HIV-1-infection
Keywords: HIV young Black men who have sex with men substance use

STUDY DESIGN:
Intervention Model Description: Mobile-enhanced engagement interventions (MEI) to support 1) HIV viral suppression among HIV-positive, not virally suppressed participants; 2) HIV-PrEP uptake among high-risk HIV-negative participants; and 3) engagement in substance abuse treatment for HIV-positive and HIV-negative participants.
Who Masked: Care Provider
Masking Description: Care providers and investigators will not know which patients are randomized to intervention or control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile-enhanced Engagement Intervention (Experimental): Mobile-enhanced engagement intervention (MEI) to support HIV-positive and high risk HIV-negative participants achieve sustained engagement and sustained retention in HIV treatment or HIV prevention (PrEP) and substance use services at 18-months.
  Interventions: Behavioral: Mobile-enhanced Engagement Intervention
- Control - SOC Case Management (No Intervention): Standard of care (SOC) case management.

INTERVENTIONS:
Behavioral: Mobile-enhanced Engagement Intervention — Mobile phone based enhanced case management intervention for HIV positive & HIV negative young Black men who have sex with men.
  Arms: Mobile-enhanced Engagement Intervention

SUMMARY:
Project Narrative This 5-city proposal seeks to address HIV disparities among young (ages 15-24) Black and/or Latinx men who have sex with men (YBLMSM) and transgender women (YBLTW) in a multilevel intervention to identify, engage and retain, high-risk HIV-uninfected and HIV-infected urban YBMSM/TW in the HIV prevention and treatment cascade. The mobile-enhanced engagement intervention (MEI) is driven by the expressed and self-determined needs of each HIV infected and uninfected participant and includes care navigation, engagement, treatment and adherence. MEI also includes a supplemental Screening, Brief Intervention, and Referral for Treatment (SBIRT), to support YBLMSM/TW who face barriers accessing substance use treatment. By building upon existing case management services and flexibility to be adapted across ages and maturity and for prevention services, this intervention has the ability to transform networks, HIV and prevention care in YBLMSM/TW in cities with very high primary and secondary HIV transmission.

DETAILED DESCRIPTION:
Project Summary The U.S. National HIV/AIDS Strategy 2020 calls for increasing access to care and improving outcomes of people living with HIV and targeting biomedical prevention efforts (including access to pre-exposure prophylaxis [PrEP]) where HIV is most heavily concentrated. Baltimore, MD; Washington, DC; Philadelphia, PA (BWP); and Tampa and St. Petersburg, FL. are disproportionately burdened by high rates of new cases of HIV infection, with disproportionate rates in young Black and/or Latinx men who have sex with men (YBLMSM) and transgender women (YBLTW) aged 15-24. High incidence underscores the need for increased identification, linkage and initiation in HIV and preventive care for YBLMSM. Grants focused on high rates directly address NIH research priorities to reduce health disparities in the incidence of HIV, in antiretroviral therapy (ART) outcomes or in high HIV prevalent or high-risk areas.

This innovative proposal seeks to test, treat and retain YBLMSM/TW living in BWP along the prevention and treatment continuum using the following aims:

Aim 1. Identify and recruit young (ages 15-24) Black and/or Latinx men who have sex with men (YBLMSM) in 3 urban cities who are (1) HIV-infected, not virally suppressed; and (2) high-risk HIV-uninfected YBLMSM, including gender variant and questioning men, using respondent driven sampling (RDS) with targeted seed identification. Assigned female sex at birth participants may be eligible to screen and participate in this aim to assist in recruiting YBLMSM/TW; Aim 2. Compare the efficacy of two study arms (mobile-enhanced engagement intervention (MEI) vs. standard of care (SOC)) to achieve sustained retention (measured by ≥ 4 follow up visits per 18-months) and engagement in HIV care (measured by durable viral suppression (HIV VL < 20 copies/ml) and substance treatment among 240 HIV-infected YBLMSM who are not virally suppressed and recruited from RDS; and Aim 3. Modify and implement mobile-enhanced intervention for 225 high-risk HIV-uninfected YBLMSM, recruited from RDS to promote linkage, retention and engagement of pre-exposure prophylaxis (PrEP) and substance treatment uptake over 18-months, comparing younger (15-19) and older (20-24) participants.

ELIGIBILITY:
Natal Male Inclusion Criteria:

* Assigned male at birth
* 15-24 years old
* English speaking
* Black/African American
* Hispanic/Latino ethnicity
* HIV positive, viral load of 20 or greater
* HIV negative, at high risk of HIV acquisition
* Sex with another male within last 12-months
* No plans to move outside of the research catchment area in next 18-months
* Able and willing to provide informed consent
* Not currently taking pre-exposure prophylaxis (PrEP)
* Not currently enrolled or planning to enrolled in an HIV vaccine trial
* Not currently enrolled or planning to enroll in an HIV adherence intervention

Natal Male Exclusion Criteria:

* Birth-identified female
* under age 15
* Over age 24
* Non-English speaking
* No sex with another male in prior 12-months
* Not Black/African American or Hispanic identified
* HIV-positive, virally suppressed
* HIV-negative, not at high risk of HIV acquisition
* Unable or unwilling to provide consent for study participation
* Unable or unwilling to return for study visits
* Unwilling to provide an oral, blood or urine specimen for testing
* Currently taking pre-exposure prophylaxis (PrEP)
* Active or previous participation in an HIV vaccine trial
* Current participation in an adherence intervention (unless proof in the non-intervention arm)
* plan to relocate out of Baltimore, Washington DC, or Philadelphia in next 18- months

Natal Female Inclusion Criteria:

* Assigned female sex at birth
* English speaking
* 15-24 years old
* Have friends who are gay or bisexual males or transgender females

Natal Female Exclusion Criteria:

* Assigned male sex at birth
* Non-English speaking
* Under age 15
* Over age 24
* No report of friends who are gay or bisexual males or transgender females

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 631 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
HIV Viral Suppression | 18-months
  Durable viral suppression (VL < 20 copies/ml)
PrEP Uptake | 18-months
  Engagement in HIV pre-exposure prophylaxis (PrEP) services

SECONDARY OUTCOMES:
Engagement in substance abuse treatment services | 6-months
  Defined as at least two substance abuse treatment visits

CONTACTS AND LOCATIONS:
Overall Officials: David Celentano, ScD, MHS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Renata Sanders, MD, ScM, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health and JHU School of Medicine
Locations (1):
- Center for Adolescent and Young Adult Health at Johns Hopkins Harriet Lane, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Arrington-Sanders R, Galai N, Falade-Nwulia O, Hammond C, Wirtz A, Beyrer C, Arteaga A, Celentano D. Patterns of Polysubstance Use in Young Black and Latinx Sexual Minority Men and Transgender Women and Its Association with Sexual Partnership Factors: The PUSH Study. Subst Use Misuse. 2024;59(3):317-328. doi: 10.1080/10826084.2023.2267655. Epub 2024 Jan 25. PMID 38146133
- [Derived] Shorrock F, Alvarenga A, Hailey-Fair K, Vickroy W, Cos T, Kwait J, Trexler C, Wirtz AL, Galai N, Beyrer C, Celentano D, Arrington-Sanders R. Dismantling Barriers and Transforming the Future of Pre-Exposure Prophylaxis Uptake in Young Black and Latinx Sexual Minority Men and Transgender Women. AIDS Patient Care STDS. 2022 May;36(5):194-203. doi: 10.1089/apc.2021.0222. PMID 35507322
- [Derived] Arrington-Sanders R, Alvarenga A, Galai N, Arscott J, Wirtz A, Carr R, Lopez A, Beyrer C, Nessen R, Celentano D. Social Determinants of Transactional Sex in a Sample of Young Black and Latinx Sexual Minority Cisgender Men and Transgender Women. J Adolesc Health. 2022 Feb;70(2):275-281. doi: 10.1016/j.jadohealth.2021.08.002. Epub 2021 Sep 24. PMID 34580030
- [Derived] Arrington-Sanders R, Hailey-Fair K, Wirtz A, Cos T, Galai N, Brooks D, Castillo M, Dowshen N, Trexler C, D'Angelo LJ, Kwait J, Beyrer C, Morgan A, Celentano D; PUSH Study. Providing Unique Support for Health Study Among Young Black and Latinx Men Who Have Sex With Men and Young Black and Latinx Transgender Women Living in 3 Urban Cities in the United States: Protocol for a Coach-Based Mobile-Enhanced Randomized Control Trial. JMIR Res Protoc. 2020 Sep 16;9(9):e17269. doi: 10.2196/17269. PMID 32935662